CLINICAL TRIAL: NCT07117747
Title: Non-invasive Skin Sampling: Optimization of Sample Collection and Extraction. Enhancing Cytokine Recovery by the Modification of Extraction Solvents and the Use of Alternative Sampling Methods
Brief Title: Non-invasive Sampling Method for Skin Test: Optimization of Sample Collection and Extraction
Acronym: SPECIMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C3351
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Absorbing hygiene product; Skin sampling; Cytokines

STUDY DESIGN:
Intervention Model Description: Samples are taken from the forearms of healthy individuals at two visits and the amount of cytokines that can be retrieved from the samples re extracted using various methods in order to optimize the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): Single arm study
  Interventions: Other: Healthy volunteers

INTERVENTIONS:
Other: Healthy volunteers — All subject belong to the same arm and ther is no intervention

SUMMARY:
When absorbent hygiene products-such as panty liners, sanitary pads, incontinence products, or wound care items-are used over extended periods, they can sometimes have negative effects on the skin. The aim of the current study is to investigate the best way to measure the amount of cytokines on the skin through a non-invasive method.

Cytokines are small proteins that act as signaling molecules in the immune system and regulate inflammation and the body's response to infections. Because inflammatory markers often appear in very low concentrations in skin surface samples, it is essential to optimize both collection and extraction methods to overcome this limitation.

The researchers want to evaluate different sampling and extraction techniques to measure the skin's inflammatory response. The effectiveness assessment involves determining how well these methods can detect and analyze inflammatory markers. This includes ensuring the sampling methods are non-invasive yet sensitive enough to detect subtle changes in skin inflammation. Furthermore, the extraction methods must efficiently isolate relevant biomarkers to provide reliable data on the skin's response to the products.

DETAILED DESCRIPTION:
The aim of this project was to refine a non-invasive skin sampling technique, enhancing cytokine recovery by optimizing both the sample collection method (tape stripping or swabbing) and the cytokine extraction solvent (including buffer type, detergent, and detergent concentration). The analytes of interest were the following five cytokines: IL-1α, IL-1RA, IL-6, IL-8, and TNF-α, which are signaling molecules in the immune system and important inflammatory biomarkers. ELISA was used for quantitative analysis.

Tape stripping and swabbing are two non-invasive skin sampling methods. For tape stripping, sample collection and extraction have been performed using D-Squame tape and an extraction buffer reported in relevant publications. Expanding the list of detectable cytokines allows for more accurate evaluations of skin condition.

ELIGIBILITY:
Inclusion Criteria:

* Sex: men/women
* Age: >18 years
* Subjects with full legal competence
* Subjects who have provided a signed informed consent and willing to come to the scheduled visit at the test site

Exclusion Criteria:

* Subjects that have participated in any skin test that could cause damage to the skin barrier during the last 2 weeks
* Subjects that have participated in any skin test that could cause damage to the skin barrier during the last 2 weeks
* Subjects with known sensitivity or allergy to adhesives and nylon
* Have immunodeficiency, taking any anti-inflammatory medication or having any other condition that makes participation in the clinical investigation inappropriate, as judged by investigator
* Subjects with hairy forearms
* Subjects with active skin diseases on the forearms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Cytokine detection | 1-2 months
  the detection of cytokines obtained by the different extraction solvents and sampling methods. ELISA complemented with the Micro BCA Protein Assay were used to quantify the cytokine recovery (in pg/ug total soluble protein).

CONTACTS AND LOCATIONS:
Overall Officials: Warangkana Lohcharoenkal, PhD, Principal Investigator — Essity Hygiene and Health AB
Locations (1):
- Essity Study Site, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No